CLINICAL TRIAL: NCT01380925
Title: Search for Novel Breast Cancer Susceptibility Genes in Pedigrees of African Ancestry
Brief Title: The Jewels in Our Genes Study - an African American Family Study of Breast Cancer
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Heather Ochs-Balcom, Assistant Professor, University at Buffalo
Other Study IDs: KG090937
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The research team is studying why some African American families have multiple cases of breast cancer.

This study will help to better understand if there are undiscovered genes unique to African Americans that may predict early breast cancer risk.

Breast cancer survivors AND their relatives who are also breast cancer survivors are being recruited to the study.

ELIGIBILITY:
Inclusion Criteria:

* Black/African American
* Ever diagnosed with breast cancer
* Have at least one living blood relative ever diagnosed with breast cancer, who is also willing to participate
* Live in the U.S.

Exclusion Criteria:

* Tested positive for BRCA mutations

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American breast cancer survivors.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ochs-Balcom HM, Sun X, Chen Y, Barnholtz-Sloan J, Erwin DO, Jandorf L, Sucheston-Campbell L, Elston RC. Putative linkage signals identified for breast cancer in African American families. Cancer Epidemiol Biomarkers Prev. 2015 Feb;24(2):442-7. doi: 10.1158/1055-9965.EPI-14-1131. Epub 2014 Dec 4. PMID 25477366